CLINICAL TRIAL: NCT04244487
Title: Vagus Nerve-preserving Laparoscopic Splenectomy and Azygoportal Disconnection With Versus Without Intraoperative Endoscopic Variceal Ligation
Brief Title: Laparoscopic Splenectomy and Azygoportal Disconnection With Intraoperative Endoscopic Variceal Ligation
Acronym: SVEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Guo-Qing Jiang, Clinical Professor, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YZUC-004
Record Dates: First submitted 2020-01-18; First posted 2020-01-28 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Cirrhosis; Hypertension; Splenectomy; Laparoscopy
Keywords: Vagus nerve; Esophageal variceal re-bleeding; Cirrhosis; Hypertension; laparoscopy
MeSH Terms: conditions — Fibrosis; Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intraoperative endoscopic variceal ligation group (Experimental): intraoperative endoscopic variceal ligation group Every patient of vagus nerve-preserving group will receive the synchronous vagus nerve-preserving laparoscopic splenectomy and azygoportal disconnection with intraoperative endoscopic variceal ligation procedure
  Interventions: Procedure: laparoscopic splenectomy and azygoportal disconnection with intraoperative endoscopic variceal ligation
- Non-intraoperative endoscopic variceal ligation group (No Intervention): Every patient of conventional group will receive single vagus nerve-preserving laparoscopic splenectomy and azygoportal disconnection without intraoperative endoscopic variceal ligation procedure

INTERVENTIONS:
Procedure: laparoscopic splenectomy and azygoportal disconnection with intraoperative endoscopic variceal ligation — The modified procedure was implemented in the following order: (1) find the left crural diaphragm; (2) via the surface of the left crural diaphragm, divide the left lateral surface of the distal esophagus; (3) divide the posterior surface of the distal esophagus; (4) divide the anterior surface of the distal esophagus; (5) divide the lesser omental sac via the bottom right crural diaphragm; (6) transect en bloc the left gastric artery and vein and posterior gastric veins using a linear laparoscopic vascular stapler; (7) find the right crural diaphragm by dividing a small portion of the hepatogastric ligament at the left lateral esophagogastric junction; and (8) via the surface of the right crural diaphragm, divide the right lateral surface of the distal esophagus.
  After the procedure of laparoscopic azygoportal disconnection, intraoperative endoscopic variceal ligation was made if the diameter of the esophageal varices was >5 mm.
  Arms: intraoperative endoscopic variceal ligation group

SUMMARY:
This study aimed to evaluate whether synchronous vagus nerve-preserving laparoscopic splenectomy and azygoportal disconnection with intraoperative endoscopic variceal ligation (SVEL) is effective and safe, and to determine whether SVEL can effectively decrease the incidence of postoperative esophageal variceal re-bleeding.

DETAILED DESCRIPTION:
After successful screening the cases of cirrhosis of liver irrespective of the etiology who have prior esophageal/gastroesophageal variceal bleeding will be enrolled. The baseline parameter will be recorded and the patient will be randomized into either interventional (synchronous vagus nerve-preserving laparoscopic splenectomy and azygoportal disconnection with intraoperative endoscopic variceal ligation (SVEL)) or control (single vagus nerve-preserving laparoscopic splenectomy and azygoportal disconnection without intraoperative endoscopic variceal ligation (SVEL)) group. From postoperative day 3, all patients will receive 100 mg oral aspirin enteric-coated tablets (Bayer, Leverkusen, Germany) once daily for 1 year, low-molecular-weight heparin (CS Bio, Hebei, China) subcutaneously (4.100 IU/day) for 5 days, and 25 mg of oral dipyridamole (Henan Furen, Henan, China) thrice daily for 3 months. At months 3, 6, and 12 after operation, endoscopic intervention will be done for all patients. Endoscopic variceal ligation was made if the diameter of the esophageal varices was >5 mm. Postoperative complications of esophageal variceal re-bleeding and death due to re-bleeding will be recorded during the postoperative first year monitoring in the both groups as per the primary or secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* A clinical, radiological or histologic diagnosis of cirrhosis of any etiology
* Splenomegaly with secondary hypersplenism
* esophageal/gastroesophageal variceal bleeding
* No evidence of portal vein system thrombosis by ultrasound evaluation and angio-CT
* Informed consent to participate in the study

Exclusion Criteria:

* Hepatocellular carcinoma or any other malignancy,
* Hypercoagulable state other than the liver disease related
* DRUGS- oral contraceptives, anticoagulation or anti-platelet drugs.
* Child - Pugh C
* Recent peptic ulcer disease
* History of Hemorrhagic stroke
* Pregnancy
* Uncontrolled Hypertension
* Age>75 yrs
* Human immunodeficiency virus (HIV) infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Esophageal variceal re-bleeding | 1 year
  Proportions of patients who will suffer from esophageal variceal re-bleeding

SECONDARY OUTCOMES:
Death due to re-bleeding | 1 year
  Proportions of patients who will suffer from death due to re-bleeding
Overall survival | 1 year
  Overall survival in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Luo-Jing Zhou, MD, Study Chair — Clinical Medical College, Yangzhou University
Locations (1):
- Clinical Medical College, Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bai DS, Jin SJ, Xiang XX, Qian JJ, Zhang C, Zhou BH, Gao TM, Jiang GQ. Vagus Nerve-Preserving Laparoscopic Splenectomy and Azygoportal Disconnection with Versus Without Intraoperative Endoscopic Variceal Ligation: a Randomized Clinical Trial. J Gastrointest Surg. 2022 Sep;26(9):1838-1845. doi: 10.1007/s11605-022-05374-1. Epub 2022 Jun 8. PMID 35676457